CLINICAL TRIAL: NCT01894477
Title: A Randomized Phase II Study of Treosulfan, Fludarabine and Low-Dose TBI as Conditioning for Allogeneic Hematopoietic Cell Transplantation in Patients With Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML)
Brief Title: Treo/Flu/TBI With Donor Stem Cell Transplant for Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joachim Deeg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2524.00; NCI-2013-01261 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2524; 2524.00 (Other: Fred Hutch/University of Washington Cancer Consortium); K12HL087165 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia in Remission; Chronic Myelomonocytic Leukemia; Minimal Residual Disease; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Neoplasm, Residual; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders | interventions — fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Arm A: Treosulfan, Fludarabine Phosphate
  Treosulfan intravenously (IV) over 2 hours on days -6 to -4 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Fludarabine Phosphate; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation; Drug: Treosulfan; Other: Laboratory Biomarker Analysis
- Arm B (Experimental): Arm B: Treosulfan, Fludarabine Phosphate, TBI
  Treosulfan and fludarabine phosphate as in Arm A and undergo low -dose total-body irradiation (TBI) on day 0
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Fludarabine Phosphate; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Treosulfan; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic bone marrow transplant
  Other Names: Allo BMT; Allogeneic BMT
Drug: Fludarabine Phosphate — Intravenously administered Fludarabine Phosphate
  Other Names: 2-F-ara-AMP; Beneflur; Fludara; SH T 586
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation
  Arms: Arm A
Drug: Treosulfan — Intravenously administered Treosulfan
  Other Names: 1,2,3, 4-Butanetetrol, 1,4-dimethanesulfonate, [R-(R*,S*)]-; Dihydroxybusulfan; Ovastat; Treosulphan; Tresulfon
Other: Laboratory Biomarker Analysis — Correlative Studies

SUMMARY:
This randomized phase II trial studies how well treosulfan and fludarabine phosphate, with or without total body irradiation before donor stem cell transplant works in treating patients with myelodysplastic syndrome or acute myeloid leukemia. Giving chemotherapy, such as treosulfan and fludarabine phosphate, and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus before and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the better of two treosulfan-based conditioning regimens in patients with myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML), by comparing 6-month progression-free survival.

SECONDARY OBJECTIVES:

I. Determine the effects of two conditioning regimens on changes in gene expression profiles, and evaluate the association of gene expression profiles and disease relapse.

II. Determine the incidence of progression-free survival at 1 year and 2 years after hematopoietic cell transplantation (HCT).

III. Evaluate overall survival (OS) at 6 months, at 1 year and at 2 years after HCT.

IV. Determine the incidence of grades II-IV acute graft-versus-host disease (GVHD).

V. Determine the incidence of chronic GVHD.

VI. Determine donor chimerism around days +28 and +84.

CONDITIONING REGIMEN:

Arm A: Patients receive treosulfan intravenously (IV) over 2 hours on days -6 to -4 and fludarabine phosphate IV over 30 minutes on days -6 to -2.

Arm B: Patients receive treosulfan and fludarabine phosphate as in Arm A and undergo low-dose total-body irradiation (TBI) on day 0.

TRANSPLANT: Patients in both arms undergo allogeneic peripheral blood stem cell (PBSC) transplant or bone marrow transplant on day 0.

GVHD PROPHYLAXIS: Patients with a related donor receive tacrolimus orally (PO) every 8 or 12 hours on days -3 to 56 with taper to day 180. Beginning 4-6 hours after PBSC infusion, patients also receive mycophenolate mofetil PO every 12 hours to day 28. Patients with an unrelated donor receive tacrolimus PO every 8 or 12 hours on days -3 to 100 with taper to day 180. Beginning 4-6 hours after PBSC infusion, patients also receive mycophenolate mofetil PO every 8 hours to day 40 with taper to day 96.

NOTE: Patients with related donors eligible for FHCRC protocol 2545 may receive cyclosporine IV, instead of tacrolimus, beginning on day -3 to day 50 with a taper to day 180.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* MDS, myelodysplastic syndrome/myeloproliferative neoplasia overlap disorders (including chronic myelomonocytic leukemia [CMML], and MDS/myeloproliferative neoplasm [MPN] unclassifiable syndromes)
* AML, other than acute promyelocytic leukemia (APL), in first or second remission or with minimal residual disease
* With Karnofsky index or Lansky Play-Performance scale > 70% on pre-transplant evaluation
* Able to give informed consent (if > 18 years), or with a legal guardian capable of giving informed consent (if < 18 years)
* Patients with previous autologous or allogeneic HCT are allowed to enroll
* DONOR: Human leukocyte antigen (HLA)-identical related donors or
* DONOR: Unrelated donors matched for HLA-A, B, C, DRB1, and DQB1 as defined by high resolution deoxyribonucleic acid (DNA) typing; mismatch for one HLA allele is allowed
* DONOR: Donors able to undergo peripheral blood stem cell collection or bone marrow harvest
* DONOR: Donors in good general health, with a Karnofsky or Lansky play performance score > 90%
* DONOR: Donors able to give informed consent (if > 18 years), or with a legal guardian capable of giving informed consent (if < 18 years)

Exclusion Criteria:

* Receiving umbilical cord blood
* With impaired cardiac function as evidenced by ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%) or cardiac insufficiency requiring treatment or symptomatic coronary artery disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* With impaired pulmonary function as evidenced by partial pressure of oxygen (pO2) < 70 mm Hg and carbon monoxide diffusing capability test (DLCO) < 70% of predicted or pO2 < 80 mm Hg and DLCO < 60% of predicted; (or, for pediatric patients unable to perform pulmonary function tests, then oxygen (O2) saturation < 92% on room air), or receiving supplementary continuous oxygen
* With impaired renal function as evidenced by creatinine-clearance < 50% for age, weight, height or serum creatinine > 2 x upper limit of normal or dialysis-dependent
* With hepatic dysfunction as evidenced by total bilirubin > 2.0 x upper limit of normal or evidence of synthetic dysfunction or severe cirrhosis
* With hepatic dysfunction as evidenced by aspartate aminotransferase (AST) > 2.0 x upper limit of normal or evidence of synthetic dysfunction or severe cirrhosis
* With active infectious disease requiring deferral of conditioning, as recommended by an infectious disease specialist
* With human immunodeficiency virus (HIV)-positivity or active infectious hepatitis
* With central nervous system (CNS) leukemic involvement not clearing with intrathecal chemotherapy, cranial irradiation or both prior to initiating conditioning (day -6)
* Patients with active non-hematological malignancies (except non-melanoma skin cancers) or those with non-hematological malignancies who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within 5 years; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* With life expectancy severely limited by diseases other than malignancy
* Women who are pregnant or lactating
* With known hypersensitivity to treosulfan or fludarabine (fludarabine phosphate)
* Receiving another experimental drug within 4 weeks before initiation of conditioning (day -6)
* Unable to give informed consent (if > 18 years) or with a legal guardian (if < 18 years) unable to give informed consent
* DONOR: Individuals deemed unable to undergo marrow harvesting or PBSC mobilization and leukapheresis
* DONOR: Individuals who are HIV-positive
* DONOR: Individuals with active infectious hepatitis
* DONOR: Females with a positive pregnancy test
* DONOR: Persons unable to give informed consent (if > 18 years) or with a legal guardian (if < 18 years) unable to give informed consent

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-11; Primary Completion 2017-01-09 (Actual); Study Completion 2022-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Treosulfan, Fludarabine Phosphate): CONDITIONING REGIMEN:
  Treosulfan IV over 2 hours on days -6 to -4 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
  TRANSPLANT: Patients in both arms undergo allogeneic PBSC transplant or bone marrow transplant on day 0.
  GVHD PROPHYLAXIS: Patients with related donor receive tacrolimus PO every 8 or 12 hours on days -3 to 56 with taper to day 180. Beginning 4-6 hours after PBSC infusion, and mycophenolate mofetil PO every 12 hours to day 28. Patients with an unrelated donor receive tacrolimus PO every 8 or 12 hours on days -3 to 100 with taper to day 180. Beginning 4-6 hours after PBSC infusion, and mycophenolate mofetil PO every 8 hours to day 40 with taper to day 96.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic bone marrow transplant
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSC
- Arm B (Treosulfan, Fludarabine Phosphate, TBI): CONDITIONING REGIMEN: Treosulfan and fludarabine phosphate as in Arm A and undergo low-dose TBI on day 0.
  TRANSPLANT: Patients in both arms undergo allogeneic PBSC transplant or bone marrow transplant on day 0.
  GVHD PROPHYLAXIS: Patients with a related donor receive tacrolimus PO every 8 or 12 hours on days -3 to 56 with taper to day 180. Beginning 4-6 hours after PBSC infusion, and mycophenolate mofetil PO every 12 hours to day 28. Patients with an unrelated donor receive tacrolimus PO every 8 or 12 hours on days -3 to 100 with taper to day 180. Beginning 4-6 hours after PBSC infusion, and mycophenolate mofetil PO every 8 hours to day 40 with taper to day 96.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic bone marrow transplant
  Fludarabine Phosphate: Given IV
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSC transplant
  Total-Body Irradation
Period: Overall Study
Arm/Group | Arm A (Treosulfan, Fludarabine Phosphate) | Arm B (Treosulfan, Fludarabine Phosphate, TBI)
Started | 35 | 67
Completed | 35 | 65
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — protocol changed due SC changed to cord | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A (Treosulfan, Fludarabine Phosphate): Treosulfan IV over 2 hours on days -6 to -4 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
- Arm B (Treosulfan, Fludarabine Phosphate, TBI): Treosulfan and fludarabine phosphate as in Arm A and undergo low-dose TBI on day 0.
- Total: Total of all reporting groups
Arm/Group | Arm A (Treosulfan, Fludarabine Phosphate) | Arm B (Treosulfan, Fludarabine Phosphate, TBI) | Total
Number analyzed (Participants) | 35 | 65 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 28 | 53 | 81
  >=65 years | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 31 | 49
  Male | 17 | 34 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 35 | 62 | 97
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 9 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 1 | 1
  White | 30 | 52 | 82
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 63 | 98
  Indonesia | 0 | 1 | 1
  Samoa | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Did Not Progress Within 6 Months
Description: Progression is defined as relapse
Time Frame: At 6 months post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Treosulfan, Fludarabine Phosphate) | Arm B (Treosulfan, Fludarabine Phosphate, TBI)
Number analyzed (Participants) | 35 | 65
Participants | 20 | 48

2. Secondary Outcome: Number of Participants With Acute GVHD, Graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: Up to 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Treosulfan, Fludarabine Phosphate) | Arm B (Treosulfan, Fludarabine Phosphate, TBI)
Number analyzed (Participants) | 35 | 65
Participants | 29 | 50

3. Secondary Outcome: Incidence of Chronic GVHD Graded by the NCI CTCAE Version 4.0
Time Frame: Up to 5 year
Reporting Status: Not Posted, anticipated posting 2023-01

4. Secondary Outcome: Incidence of Relapse/Progression
Time Frame: Up to 5 year
Reporting Status: Not Posted

5. Secondary Outcome: NRM
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 2 year
Reporting Status: Not Posted

7. Secondary Outcome: Change in Gene Expression Profiles
Description: Differences between arms in the changes in gene expression will be compared. 80% power to detect mean differences of approximately 1.4 standard deviation units, at the 2-sided 0.05 level of significance (with Bonferroni correction for 50 genes).
Time Frame: Baseline and at day 0 within 6 hours of conditioning prior to transplant
Reporting Status: Not Posted, anticipated posting 2022-06

8. Secondary Outcome: Relapse Risk as Measured by Degree of Change in Gene Expression Profiles
Description: Among genes identified whose expression is modified by conditioning, degree of change in expression will be evaluated to determine if it is correlated with relapse risk and offers improved prediction of relapse risk over that obtained with standard clinical parameters (cytogenetics, blast count, International Prognostic Scoring System score, minimal residual disease. To account for censoring and the competing risk of non-relapse mortality (NRM), the analysis will be a time-to-event analysis of relapse using Cox regression, with change in expression as a continuous covariate (on a log scale). 8
Time Frame: Baseline and at day 0 within 6 hours of conditioning prior to transplant
Reporting Status: Not Posted, anticipated posting 2022-06

ADVERSE EVENTS:
Time Frame: Regimen-related toxicity and infection will be evaluated up to the time the patient is discharged from medical care at the transplant institution, or day 100.
Description: Regimen-related toxicity, greater or equal to grade 3, excluding cytopenias, and infection will be evaluated up to the time the patient is discharged from medical care at the transplant institution, or day 100. Toxicities will be documented per Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
  All patients undergoing HCT are expected to have Grade 3 and 4 pancytopenia as an intended therapeutic effect, and thus this will not be reported as an adverse event.
Arm/Group | Arm A (Treosulfan, Fludarabine Phosphate) | Arm B (Treosulfan, Fludarabine Phosphate, TBI)
All-Cause Mortality (participants affected / at risk) | 15/35 | 20/67
Serious Adverse Events (participants affected / at risk) | 6/35 | 9/67
Other Adverse Events (participants affected / at risk) | 28/35 | 51/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Treosulfan, Fludarabine Phosphate) (N=35) | Arm B (Treosulfan, Fludarabine Phosphate, TBI) (N=67)
GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
CMV Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
loss of vision (Eye disorders) | 1 (1) | 0 (0)
Engraftment syndrome (Immune system disorders) | 1 (1) | 0 (0)
mental status changes (Psychiatric disorders) | 2 (2) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post Transplant Lymphoproliferative Disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Total body edema (General disorders) | 1 (1) | 0 (0)
Steroid myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Treosulfan, Fludarabine Phosphate) (N=35) | Arm B (Treosulfan, Fludarabine Phosphate, TBI) (N=67)
Atrial fibrillation/flutter (Cardiac disorders) | 0 (0) | 3 (3)
Decreased LVEF (Cardiac disorders) | 0 (0) | 2 (2)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Elevated BNP (Cardiac disorders) | 0 (0) | 1 (1)
Deconditioned (General disorders) | 3 (3) | 2 (2)
Edema (General disorders) | 2 (2) | 1 (1)
Fluid overload (General disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6) | 14 (14)
Vomiting (Gastrointestinal disorders) | 7 (7) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Anorexia (Gastrointestinal disorders) | 4 (4) | 7 (7)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
mucositis (Gastrointestinal disorders) | 1 (1) | 5 (5)
Typhilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated total bilirubin (Hepatobiliary disorders) | 1 (1) | 2 (2)
Elevated Alanine transaminase (Hepatobiliary disorders) | 1 (1) | 0 (0)
sinusoidal obstruction syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) — Veno-occlusive disease
Engraftment syndrome (Immune system disorders) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 20 (35) | 33 (54) — Includes bacterial, viral, and fungal
Steroid myopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7) — Includes limb, neck or back pain.
Myalgia/Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Septic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminenia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 9 (9)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Posttransplant lymphoproliferative disease (PTLD-DLBC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
mental status changes (Psychiatric disorders) | 1 (1) | 3 (3)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasms (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Peeling blisters (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes